CLINICAL TRIAL: NCT02908048
Title: Extracellular RNA Markers of Liver Disease and Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tushar Patel, Professor, Mayo Clinic
Other Study IDs: 14-004560
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma; Biliary Tract Cancer; Cirrhosis; Liver Diseases
Keywords: liver cancer; cholangiocarcinoma (CCA); cirrhosis; hepatitis; bile duct cancer; hepatocellular carcinoma (HCC); hepatobiliary carcinoma; hepatoma; liver mass
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms; Fibrosis; Liver Diseases; Liver Neoplasms; Cholangiocarcinoma; Hepatitis; Bile Duct Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hepatocellular Carcinoma: Blood samples will be collected at entry into the study and at varying intervals over a two to three year period.
  Interventions: Other: Blood samples
- Biliary Tract Cancer: Blood samples will be collected at entry into the system and at varying intervals over a two to three year period.
  Interventions: Other: Blood samples
- Cirrhosis: Blood samples will be collected during regular intervals over a three year period.
  Interventions: Other: Blood samples
- Chronic Liver Disease without Cirrhosis: A single blood sample will be collected at entry into the study
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples collected at varying intervals over a two to three year period.

SUMMARY:
The study will examine and evaluate the use of extracellular RNA in blood as markers for the diagnosis of liver disease or cancer, and as markers for prediction of response to treatment or recurrence of cancer after surgery

DETAILED DESCRIPTION:
The goal is to identify an extracellular RNA candidate for the detection and diagnosis of liver cancers such as hepatocellular cancer or biliary cancer, and chronic liver diseases. The use of selected exRNA biomarkers for diagnosis of hepatocellular cancer (HCC) or biliary tract cancers in patients with cirrhosis will be evaluated in a prospective case-control study. The study will create a registry of patients who have chronic liver disease, cirrhosis, liver and biliary tract cancers. A risk factor questionnaire will be administered to facilitate identification of risk factors for development of liver cancer. Patient information will be obtained from the medical record, and include demographics, medical history, liver disease, smoking and alcohol history, etiology, family history, and clinical laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* Lab results from within the previous 90 days.
* Diagnosis of HCC or biliary tract cancer
* Diagnosis of cirrhosis based on histology, imaging, or ultrasound.
* Diagnosis of a chronic liver disease without cirrhosis.

Exclusion Criteria for the HCC/biliary tract cancer group:

* Prior solid organ transplant.
* Previous cancer history with the last 5 years (excluding non-melanoma skin cancer), participation in a treatment trial for HCC

Exclusion criteria for the cirrhosis and chronic liver disease groups:

* Prior solid organ transplant.
* Previous or current cancer history within the past 5 years (excluding non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing evaluation at Mayo Clinic Florida Liver Transplant, Surgery, Oncology or Radiology clinics who have hepatocellular carcinoma (HCC) or biliary tract cancers, cirrhosis without HCC, or chronic liver disease without cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 1810 (Actual)
Dates: Start 2014-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of liver cancer based on tumor markers and imaging studies. | Five years
  The exRNA biomarker levels in the HCC and biliary tract cancer groups will be evaluated and compared to the exRNA biomarker levels present in the case-control groups, cirrhosis and chronic liver disease. Statistical analysis will be used to evaluate the sensitivity and specificity of these markers for the diagnosis of cancers based on findings of liver mass, imaging characteristics, size, and extent of viable tumor on imaging, or on elevated levels of tumor markers such as alphafetoprotein.

CONTACTS AND LOCATIONS:
Overall Officials: Tushar Patel, MBChB, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Florida, Jacksonville, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - McGuire VA Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials